CLINICAL TRIAL: NCT02359669
Title: Effect of a Nutritional Approach in Combination With Cognitive Stimulation on Child Cognitive Abilities
Acronym: Stimulearn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 13.11NRC
Record Dates: First submitted 2015-01-26; First posted 2015-02-10 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2015-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Growing up milk (GUM) (Active Comparator): GUM associated with StimuLearn intervention.
  Interventions: Behavioral: StimuLearn Intervention
- Skimmed Milk (Placebo Comparator): Control group given skimmed milk without StimuLearn intervention.
  Interventions: Behavioral: Without StimuLearn intervention

INTERVENTIONS:
Behavioral: StimuLearn Intervention — * StimuLearn apps
  * Cognitive questionnaires
  Arms: Growing up milk (GUM)
Behavioral: Without StimuLearn intervention — Cognitive Questionnaires
  Arms: Skimmed Milk

SUMMARY:
The objective of the study is to explore the impact of a combined intervention including a growing up milk (GUM) fortified in micronutrients and cognitive stimulation on cognitive abilities, mother-child- interaction and behavior in children of 3 to 5 years from less enriched home environments.

DETAILED DESCRIPTION:
The objective of the study is to explore the impact of a combined intervention including a growing up milk (GUM) fortified in micronutrients and cognitive stimulation on cognitive abilities, mother-child- interaction and behavior in children of 3 to 5 years from less enriched home environments with HOME score less than 26. The control group will receive skimmed milk but no extra stimulation materials ( however, no restrictions on normal mother-child interaction). The cognitive abilities, mother-child interaction and child behavior will be assessed after a 6 months intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female children, age 3;0-4;11 years
* Having obtained their legal representative's informed consent
* Level of stimulation in their home environment score below 26 in HOME inventory
* Normal cognitive development

Exclusion Criteria:

* Neurological disorders
* Food allergies (especially milk and soy allergy)
* Documented lactose intolerance
* Children with special nutritional needs
* Children under chronic (more than 7 consecutive days) medications which may impact cognitive performance
* Children not living in a family/children in foster homes
* Subject who cannot be expected to comply with study procedures
* Currently participating or having participated in another clinical study during the last 4 weeks prior to the beginning of this study

Ages: 36 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Cognitive abilities using Wechsler Pre-School and Primary Scale of Intelligence (WPPSI-IV), 4th Edition. | 24 weeks
  Blind assessment achieved by dedicated pyschologists at test center through use of the Wechsler Pre-School and Primary Scale of Intelligence (WPPSI-IV), 4th Edition questionnaire. This test is aimed at measuring overall cognitive abilities.

SECONDARY OUTCOMES:
Parent-rating of child's development | 24 weeks.
  Measured by the Ages & Stages Questionnaire ( ASQ-3) which is a questionnaire for different age stages between 2 and 66 months of age to screen areas of communication, gross motor, fine motor, problem-solving and personal-social skills.
Mother-Child interaction | 24 weeks
  Interaction is videotaped for 10 minutes sequences and analyzed using the Parenting Interactions with Children: Checklist of Observations Linked to Outcomes (PICCOLO).
Child Behavior assessed by Child Behavior Checklist (CBCL 1.5 - 5 years) | 24 weeks
  This is a parent rated scale that obtains information about young children behaviors and is applicable for children aged 1.5 - 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Sudigdo Sastroasmoro, M.D, Ph.D, Principal Investigator — Center for Clinical Epidemiology and Evidence-based Medicine, Medical School, University of Indonesia-RSCM Hospital
Locations (1):
- Center for Clinical Epidemiology and Evidence-Based Medicine, University of Indonesia-RSCM Hospital, Jarkarta, Jarkarta, Indonesia

REFERENCES:
- [Derived] Schneider N, Geiser E, Gosoniu LM, Wibowo Y, Gentile-Rapinett G, Tedjasaputra MS, Sastroasmoro S. A Combined Dietary and Cognitive Intervention in 3(-)5-Year-Old Children in Indonesia: A Randomized Controlled Trial. Nutrients. 2018 Oct 1;10(10):1394. doi: 10.3390/nu10101394. PMID 30275398